CLINICAL TRIAL: NCT05653726
Title: Impact of Noninvasive Telemonitoring on Clinical Events, Healthcare Resource Use and Costs in Heart Failure
Brief Title: Multidimensional Impact of Telemonitoring in Heart Failure (IMPACT-HF)
Acronym: IMPACT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Fundacion Investigacion Biomedica Hospital 12 de Octubre (Unknown); Hospital Universitario Puerta de Hierro de Majadahonda (Unknown)
Responsible Party: Principal Investigator, Juan Carlos López-Azor, Principal Investigator, Doctor in Medicine, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HU12Octubre
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemonitoring group (Experimental): Follow-up group by telematic consultations and non-invasive daily telemonitoring of weight, blood pressure, heart rate, peripheral oxygen saturation and electrocardiogram.
  Interventions: Other: Telemonitoring follow-up using medical devices and telematic consultations
- Control gropu (No Intervention): Usual care follow-up group

INTERVENTIONS:
Other: Telemonitoring follow-up using medical devices and telematic consultations — Home telemonitoring of blood pressure, heart rate and peripheral oxygen saturation on a daily basis during 12 months
  Arms: Telemonitoring group

SUMMARY:
The goal of this clinical trial is to know if telemonitoring and telematic follow-up reduces the healthcare resources utilization, healthcare costs and non-healthcare costs of patients with high-risk heart failure. The main questions it aims to answer are:

* Does telematic follow-up reduce de use of healthcare resource utilization of patients with heart failure?
* Is telematic follow-up cost-efficient in terms of reducing direct healthcare costs in heart failure patients?
* Is telematic follow-up cost-efficient in terms of reducing non-healthcare costs in heart failure patients? Participants will be randomized to usual care (control group) or telematic care (interventional group). Patients randomized to the interventional group will be included in a protocol of daily automatic telemonitoring of arterial pressure, peripheral oximetry, heart rate and weight, and telematic consultations lead by a heart failure clinical specialized team.

Researchers will compare the healthcare resource utilization, healthcare and non-healthcare costs of patients randomized to control vs. interventional group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HF according to the 2021 guidelines of the European Society of Cardiology criteria for ≥3 months.
* Admitted for decompensation of chronic HF.
* Admitted for HF decompensation ≥30 days and ≤6 months.
* HF decompensation in ≥30 days and ≤6 months but discharged directly from the emergency department or managed on an outpatient basis, but requiring intravenous diuretic administration in an ambulatory basis, or >50% increase in loop diuretic dose.
* With previous optimized prognostic medical treatment.
* Under treatment with loop diuretic drugs.
* New York Heart Association functional class II, III or IV.

Exclusion Criteria:

* Inclusion in other intervention studies.
* Hemodynamic instability.
* Acute myocardial infarction, acute pulmonary thromboembolism or stroke in the previous 40 days.
* Uncontrolled arrhythmias
* On waiting list for transplantation (any organ) or other cardiac surgery.
* Advanced mechanical circulatory support.
* Chronic renal disease on hemodialysis.
* Life expectancy less than 1 year.
* Moderate-severe cognitive impairment.
* Manifest inability to use a technological system.
* Institutionalized.
* Limiting psychiatric pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health care costs | 12 months
  Sum of the costs for the consumption of medicines, primary care consultations, specialist consultations, hospitalization, emergency care and medical transport.

SECONDARY OUTCOMES:
Non-health care costs | 12 months
  Sum of informal costs (care provided by people who are not health or social care professionals) and professional costs (home help, tele-health, tele-assistance, ambulatory care centers and use of nursing homes)
Symptoms | 12 months
  Measured using New York Heart Association dyspnea scale
Care burden of caregivers | 12 months
  Measured using Zarit scale (values 0 to 88)
Number of hospital admissions | 12 months
  For any cause, cardiovascular and for heart failure.
Mortality | 12 months
  For any cause and for cardiovascular cause
Patient satisfaction with service | 12 months
  Measured using a customer satistaction questionnaire (values 0 to 20), with higer scores meaning
Adherence to the telemonitoring protocolo | 12 months
  Number of transmissions made versus planned at 12 months.
Quality of life variation | 12 months
  Euroqol-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No